CLINICAL TRIAL: NCT06317948
Title: Improving the Quality of Radiotherapy by Multi-Institution Knowledge-Based Planning Optimization Models
Brief Title: Improving the Quality of Radiotherapy by Multi-Institution Knowledge-Based Planning Optimization Models (Acronym: MIKAPOCo, Multi-Institutional Knowledge-based Approach in Plan Optimization for the Community)
Acronym: MIKAPOCo
Status: Enrolling by invitation | Type: Observational
Sponsor: IRCCS Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Claudio Fiorino, Principal Investigator, IRCCS Ospedale San Raffaele
Other Study IDs: IG23150
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer; Prostate Cancer
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: treatment plan comparison — In order to assess inter-Institute variability of DVH prediction of the various models, for the different situations and the different OARs, DVH and dose statistics (min, mean, median, max and SD of the dose received by each OAR) predicted on the patients owning to the different centers by the different models will be compared

SUMMARY:
Investigators central hypothesis is that it is possible to create libraries of "consistent" Knowledge-Based plan-models derived from large Institutional experiences. These libraries can be used to guide automated RT planning and serve as tools to assist centers for plan quality assurance (QA) and plan prediction.

Quantifying Inter-institute variability of RT planning and building libraries of interchangeable and validated multi-Institutional KB plan prediction models is expected to impact on the quality of planning at the national level. The project has the potential of facilitating the introduction of AI approaches in plan optimization, thus reducing intra and inter-Institute planning variability. Improving plan quality is expected to translate into better outcome after RT in terms of local control and, even more, of side effects and Quality of life. Positive impact is also expected in patient selection for advanced techniques, in plan audit and plan optimization in clinical trials, in technology comparison and cost-benefit analyses as well as in the RT educational field.

DETAILED DESCRIPTION:
Major aims

1. To create libraries of consistently generated KB models for patients treated with RT for breast and prostate cancer and for selected stereotactic-body RT (SBRT) applications based on the experience of many Italian Institutions; to quantify planning inter-institute variability in homogeneous classes of patients.
2. To group models based on their characteristics and interchangeability. To assess groups of highly interchangeable models to be considered for multi-institutional dose-volume histogram (DVH) prediction purposes.

ELIGIBILITY:
Inclusion Criteria:

* real life consecutive (or randomly chosen) plan data of patients treated for prostate cancer during the last 10 years;
* real life consecutive (or randomly chosen) plan data of patients treated for breast cancer during the last 10 years;
* real life consecutive (or randomly chosen) plan data of patients treated for selected SBRT situations (spine and prostate, according to RTOG 0631 and 0938 schemes respectively) during the last 10 years.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: prostate cancer, breast cancer and for selected SBRT situations (spine and prostate, according to RTOG 0631 and 0938 schemes respectively).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-10-28 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2025-10-28 (Estimated)

PRIMARY OUTCOMES:
model interchangeability | 3 years
  interchangeability will be assessed by considering: a) the fraction of patients identified as "anatomy outlier" (in terms of out of the geometric features (GF) boundary of each single model) once the model coming from Institute X is applied to patients of Institute Y (modX-Y) and vice-versa (modY-X); b) the relative differences in DVH predictions between modX-Y and modY-X, including and not including the previously recognized "GF outlier" patients. Based on these results and on their clinical interpretation, sub-groups of KB-models with "high" interchangeability will be tentatively identified and the relationships between GF and interchangeability quantified.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Fiorino, Msc, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Esposito PG, Castriconi R, Mangili P, Broggi S, Fodor A, Pasetti M, Tudda A, Di Muzio NG, Del Vecchio A, Fiorino C. Knowledge-based automatic plan optimization for left-sided whole breast tomotherapy. Phys Imaging Radiat Oncol. 2022 Jun 23;23:54-59. doi: 10.1016/j.phro.2022.06.009. eCollection 2022 Jul. PMID 35814259
- [Background] Tudda A, Castriconi R, Benecchi G, Cagni E, Cicchetti A, Dusi F, Esposito PG, Guernieri M, Ianiro A, Landoni V, Mazzilli A, Moretti E, Oliviero C, Placidi L, Rambaldi Guidasci G, Rancati T, Scaggion A, Trojani V, Fiorino C. Knowledge-based multi-institution plan prediction of whole breast irradiation with tangential fields. Radiother Oncol. 2022 Oct;175:10-16. doi: 10.1016/j.radonc.2022.07.012. Epub 2022 Jul 19. PMID 35868603
- [Background] Monticelli D, Castriconi R, Tudda A, Fodor A, Deantoni C, Gisella Di Muzio N, Mangili P, Del Vecchio A, Fiorino C, Broggi S. Knowledge-based plan optimization for prostate SBRT delivered with CyberKnife according to RTOG0938 protocol. Phys Med. 2023 Jun;110:102606. doi: 10.1016/j.ejmp.2023.102606. Epub 2023 May 15. PMID 37196603
- [Background] Castriconi R, Esposito PG, Tudda A, Mangili P, Broggi S, Fodor A, Deantoni CL, Longobardi B, Pasetti M, Perna L, Del Vecchio A, Di Muzio NG, Fiorino C. Replacing Manual Planning of Whole Breast Irradiation With Knowledge-Based Automatic Optimization by Virtual Tangential-Fields Arc Therapy. Front Oncol. 2021 Aug 24;11:712423. doi: 10.3389/fonc.2021.712423. eCollection 2021. PMID 34504790
- [Derived] Placidi L, Griffin P, Castriconi R, Tudda A, Benecchi G, Burns M, Cagni E, Markham C, Landoni V, Moretti E, Oliviero C, Guidasci GR, Meffe G, Rancati T, Scaggion A, McGoldrick K, Panettieri V, Fiorino C. An International Inter-Consortium Validation of Knowledge-Based Plan Prediction Modeling for Whole Breast Radiotherapy Treatment. Cancers (Basel). 2025 Nov 5;17(21):3576. doi: 10.3390/cancers17213576. PMID 41228368